CLINICAL TRIAL: NCT01954082
Title: INS-3: A Phase 3, Randomized, Double-Masked, Placebo-Controlled Study of the Efficacy and Safety of Myo-Inositol 5% Injection to Increase Survival Without Severe Retinopathy of Prematurity (Reduce-ROP) in Extremely Premature Infants
Brief Title: Inositol to Reduce Retinopathy of Prematurity
Acronym: INS-3
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated due to safety concerns; participant follow up will continue until March 2018
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Eye Institute (NEI) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NICHD-NRN-0053; U10HD021364 (NIH); U10HD040689 (NIH); U10HD021385 (NIH); U10HD027851 (NIH); U10HD027853 (NIH); U10HD027856 (NIH); U10HD027904 (NIH); U10HD027880 (NIH); U10HD034216 (NIH); U10HD021373 (NIH); U10HD040492 (NIH); U10HD053109 (NIH); U10HD053089 (NIH); U10HD068244 (NIH); U10HD068263 (NIH); U10HD068270 (NIH); U10HD068278 (NIH); U10HD068284 (NIH); U10HD036790 (NIH)
Record Dates: First submitted 2013-09-26; First posted 2013-10-01 (Estimated); Results first posted 2018-09-26 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Retinopathy of Prematurity (ROP)
Keywords: Retinopathy; Prematurity; Infant, Newborn, Diseases
MeSH Terms: conditions — Retinopathy of Prematurity; Retinal Diseases; Premature Birth; Infant, Newborn, Diseases | interventions — Inositol; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- myo-Inositol 5% Injection (Experimental): Within 12-72 hours of birth, infants will receive 80 mg myo-inositol 5% Injection per kilogram per day, administered in divided doses every 12 hours (40 mg/kg/dose). Study drug will be administered daily and continued until the earliest of 34 completed weeks PMA, 10 weeks (70 days) chronologic age, or the time of discharge. myo-Inositol 5% Injection will be administered IV until enteral feedings are established, at which time the same dose and formulation will be administered enterally every 12 hours.
  Interventions: Drug: myo-Inositol 5% Injection
- 5% glucose(dextrose) (Placebo Comparator): Within 12-72 hours of birth, infants will receive 80 mg 5% glucose(dextrose) USP for intravenous infusion per kilogram per day, administered in divided doses every 12 hours (40 mg/kg/dose). Study drug will be administered daily and continued until the earliest of 34 completed weeks PMA, 10 weeks (70 days) chronologic age, or the time of discharge. myo-Inositol 5% Injection will be administered IV until enteral feedings are established, at which time the same dose and formulation will be administered enterally every 12 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: myo-Inositol 5% Injection — Abbott Nutrition Division, Abbott Laboratories is supplying myo-Inositol 5% Injection to the clinical centers for the duration of the trial.
  Inositol: myo-Inositol 5% Injection is an isotonic, preservative-free, sterile 5% solution of myo-inositol in water containing 0.5 gm sodium chloride per liter (8.55mM), pH 6.5-7.5. It is administered via IV infusion using syringe pump over 15-30 minutes twice per day at 12-hour intervals at a dose of 80 mg inositol/kg/day (40 mg inositol/kg/dose), which is equivalent to 1.6 mL/kg/day (0.80 mL/kg/dose).
  Other Names: Inositol
  Arms: myo-Inositol 5% Injection
Drug: Placebo — % glucose(dextrose)
  Arms: 5% glucose(dextrose)

SUMMARY:
This is a Phase 3, randomized, double-masked, placebo-controlled study designed to determine the effectiveness of myo-Inositol 5% Injection to increase the incidence of survival without severe Retinopathy of Prematurity (ROP) through acute/final ROP determination up to 55 weeks postmenstrual age (PMA) in premature infants <28 0/7 weeks' gestation.

DETAILED DESCRIPTION:
Approximately 1760 infants are to be enrolled at approximately 18 Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Neonatal Research Network (NRN) Centers (approximately 44 sites) in the United States. Infants meeting the study selection criteria and for whom informed consent is obtained will be randomized to receive either 80 mg inositol/kg/day or placebo, administered in divided doses every 12 hours (40 mg/kg/dose). Study drug will be administered daily, starting within 12 to 72 hours of birth and continued until the earliest of 34 weeks PMA, 10 weeks chronologic age, or the time of hospital discharge or transfer. Inositol or placebo will be administered IV until enteral feedings reach 120ml/kg/day (or sooner if the infant is no longer receiving IV fluids), at which time the same dose and formulation will be administered enterally every 12 hours.

For publication purposes, the analysis of the primary efficacy outcome will consider the entire study population. In support of a new drug application (NDA) for use of myo-Inositol 5% Injection to increase survival without severe ROP through the determination of acute/final ROP status, the analysis of the primary efficacy outcome will be conducted for the entire study population and separately within pre-specified regulatory sub-studies created by administratively splitting infants enrolled at each study center into two sub-studies.

Assessments performed during the study include customary newborn intensive care procedures including repeat eye examinations until ROP status is final (which often extends after discharge), measurements of growth, cranial ultrasounds or other imaging per usual practice, and the collection of clinical diagnoses throughout hospitalization to evaluate other common morbidities of extreme preterm birth. Adverse events will be recorded from time of treatment initiation until 7 days after the last dose of study drug, and concurrent medications will be recorded from 24 hours prior to randomization until 7 days after the last dose of study drug or until discharge or transfer if sooner. Using the separate NICHD Follow-up protocol, longer term data will be collected at 22-26 months corrected age, including growth, neurodevelopmental testing, overall health status, rehospitalizations, surgeries and diagnoses, including ophthalmic diagnoses and treatments since discharge.

ELIGIBILITY:
Inclusion Criteria:

* Inborn or out born infants of either gender or any race with best obstetrical estimate of gestation <28 weeks (27 6/7 weeks and younger). Gestational age will be determined by best obstetrical estimate using the hierarchy of best obstetrical estimate using early ultrasound dating, maternal menstrual dating confirmed by examination, or neonatal gestational age assessment by physical examination.
* Alive at 12 hours.
* Age in hours up to 72 hours, although we will seek enrollment as early as feasible after consent and 12 hours.
* Informed consent signed and dated by parent and/or guardian, which includes likelihood of completing follow-up ophthalmic examinations as an outpatient, and long-term follow-up.

Exclusion Criteria

* Major congenital malformations
* Congenital malformations of the eye identified prior to randomization.
* Overt evidence of intrauterine congenital infections ("TORCH") or life threatening impairment of renal, hepatic, or cardiac function (considered moribund).

Ages: 12 Hours to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 638 (Actual)
Dates: Start 2014-04-17; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele C Walsh, MD, Principal Investigator — Case Western Reserve University, Rainbow Babies and Children's Hospital; Abhik Das, PhD, Principal Investigator — RTI International; Seetha Shankaran, MD, Principal Investigator — Wayne State University; Barbara J Stoll, MD, Principal Investigator — Emory University; Kurt Schibler, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Greg Sokol, MD, Principal Investigator — Indiana University; Abbot R Laptook, MD, Principal Investigator — Brown University, Women & Infants Hospital of Rhode Island; Krisa P Van Meurs, MD, Principal Investigator — Stanford University; Waldemar A Carlo, MD, Principal Investigator — University of Alabama at Birmingham; Kathleen A Kennedy, MD, MPH, Principal Investigator — The University of Texas Health Science Center, Houston; Ronald N Goldberg, MD, Principal Investigator — Duke University; Edward F Bell, MD, Principal Investigator — University of Iowa; Dale L Phelps, MD, Study Director — University of Rochester; Carl T D'Angio, MD, Principal Investigator — University of Rochester; William Truog, MD, Principal Investigator — Children's Mercy Hospital Kansas City; Pablo Sanchez, MD, Principal Investigator — Research Institute at Nationwide Children's Hospital; Uday Devaskar, MD, Principal Investigator — University of California, Los Angeles; Myra Wyckoff, MD, Principal Investigator — University of Texas at Southwestern; Kristi L Watterberg, MD, Principal Investigator — University of New Mexico; Barbara Schmidt, MD, Principal Investigator — University of Pennsylvania
Locations (19):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California - Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Wayne State University, Detroit, Michigan
  - Children's Mercy Hospital, Kansas City, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - RTI International, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - Univeristy of Pennsylvania, Philadelphia, Pennsylvania
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
NIH has had a long-standing policy to share and make available to the public the results and accomplishments of the activities that it funds. The NRN plans to share de-identified data after final publication in an NIH supported data repository such as the NICHD Data and Specimen Hub (https://dash.nichd.nih.gov).
Supporting Information: Study Protocol
Time Frame: One year after primary publication
Access Criteria: NICHD Data and Specimen Repository (DASH)
URL: https://dash.nichd.nih.gov/

REFERENCES:
- [Derived] Brumbaugh JE, Bell EF, Hirsch SC, Crenshaw EG, DeMauro SB, Adams-Chapman IS, Lowe JR, Natarajan G, Wyckoff MH, Vohr BR, Colaizy TT, Harmon HM, Watterberg KL, Hintz SR; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Relationships between retinopathy of prematurity without ophthalmologic intervention and neurodevelopment and vision at 2 years. Pediatr Res. 2023 Nov;94(5):1720-1730. doi: 10.1038/s41390-021-01778-y. Epub 2021 Oct 22. PMID 34686832
- See also: NICHD NRN Website — http://neonatal.rti.org/
- See also: NICHD Pregnancy & Perinatology Branch — https://www.nichd.nih.gov/about/org/der/branches/ppb/Pages/projects.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From April 2014 to September 2015, infants born before 28 weeks gestation and surviving >12 hours were screened when admitted to one of the 18 NICHD NRN Centers (approximately 44 sites) in the United States and enrolled in the study if they met the eligibility criteria and consent was obtained before 72 hours postnatal age.
Groups:
- Myo-Inositol 5% Injection: Inositol (i.e myo-Inositol) 5% Injection is an isotonic, preservative-free, sterile 5% solution of myo-inositol in water containing 0.5 gm sodium chloride per liter (8.55mM), pH 6.5-7.5. The medication is administered twice per day at 12-hour intervals at a dose of 80 mg inositol/kg/day (40 mg inositol/kg/dose), which is equivalent to 1.6 mL/kg/day (0.80 mL/kg/dose) begining within 12-72 hours of birth and continuing until the earliest of 34 weeks postmenstrual age (PMA), 10 weeks chronologic age, or the time of discharge. The doses are administered intravenously (IV) using syringe pump over 15-30 minutes until enteral feeds reach 120ml/kg/day (or sooner if the infant is no longer receiving IV fluids), at which time the same dose and formulation will be administered enterally.
- 5% Glucose(Dextrose): The placebo is 5% dextrose (5% glucose) in sterile water (D5W pyrogen and preservative free) United States Pharmacopoeia (USP) for IV infusion. The placebo is administered in the same dose (80 mg glucose/kg/day divided in 2 doses administered every 12 hours) and dispensed in the same manner (intravenously or enterally) as the inositol.
Period: Overall Study
Arm/Group | Myo-Inositol 5% Injection | 5% Glucose(Dextrose)
Started | 317 | 321
Treated | 313 (The 4 participants who were not treated either died (3) or withdrew before treatment start (1).) | 319 (The 2 participants who were not treated died before treatment start.)
Completed | 249 (There were 22 infants that received more doses than intended per protocol.) | 264 (There were 27 infants that received more doses than intended per protocol.)
Not Completed | 68 | 57
Not completed — Study Suspension | 42 | 36
Not completed — Adverse Event | 10 | 4
Not completed — Intolerance | 0 | 1
Not completed — Non-compliance | 6 | 4
Not completed — Physician Decision | 2 | 0
Not completed — Parent Decision | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Discontinued Early Prior to Transfer | 3 | 2
Not completed — Redirection of Care | 0 | 2
Not completed — Miscalculation of Final Dose Day | 0 | 3
Not completed — Comfort Care | 0 | 1
Not completed — Infant Moved | 0 | 1
Not completed — Randomized not Treated | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Myo-Inositol 5% Injection | 5% Glucose(Dextrose) | Total
Number analyzed (Participants) | 317 | 321 | 638
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 25.64 (1.42) | 25.72 (1.34) | 25.68 (1.38)
Age, Continuous [Median (Full Range); unit: weeks] | 25.9 [22.0 to 27.9] | 25.9 [22.7 to 27.9] | 25.9 [22.0 to 27.9]
Age, Customized [Count of Participants; unit: Participants]
  Gestational Age: <26 weeks | 169 | 170 | 339
  Gestational Age: >=26 weeks | 148 | 151 | 299
Age, Customized [Mean (Standard Deviation); unit: Days] — Population: Age at start of study therapy is only available for infants who started treatment (313 Inositol and 319 Placebo).
  Days
    AGE AT START OF STUDY THERAPY: number analyzed (Participants) | 313 | 319 | 632
    AGE AT START OF STUDY THERAPY | 2.8 (0.8) | 2.8 (0.8) | 2.8 (0.8)
Age, Customized [Median (Full Range); unit: Days] — Population: Age at start of study therapy is only available for infants who started treatment (313 Inositol and 319 Placebo).
  Days
    AGE AT START OF STUDY THERAPY: number analyzed (Participants) | 313 | 319 | 632
    AGE AT START OF STUDY THERAPY | 3 [1 to 5] | 3 [1 to 7] | 3 [1 to 7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159 | 158 | 317
  Male | 158 | 163 | 321
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Asian | 11 | 6 | 17
  Race/Ethnicity: Black Not Hispanic or Latino | 119 | 113 | 232
  Race/Ethnicity: Hispanic or Latino | 38 | 45 | 83
  Race/Ethnicity: Other | 3 | 11 | 14
  Race/Ethnicity: White Not Hispanic or Latino | 133 | 132 | 265
  Race/Ethnicity: Unknown/Not Reported | 13 | 14 | 27
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 317 | 321 | 638
BIRTH WEIGHT [Mean (Standard Deviation); unit: Grams] | 776.1 (195) | 784.6 (198.2) | 780.4 (196.5)
BIRTH WEIGHT [Median (Full Range); unit: Grams] | 740 [394 to 1390] | 765 [300 to 1589] | 750 [300 to 1589]
ANTENATAL STEROIDS [Count of Participants; unit: Participants]
  No | 36 | 37 | 73
  Yes | 281 | 283 | 564
  Unknown/Not Reported | 0 | 1 | 1
EARLY ONSET SEPSIS [Count of Participants; unit: Participants]
  No | 310 | 312 | 622
  Yes | 7 | 9 | 16
APGAR-5 MINUTE [Count of Participants; unit: Participants]
  Test Result Available | 313 | 316 | 629
  Test Result Not Available | 4 | 5 | 9
APGAR-5 MINUTE [Median (Full Range); unit: Units on a Scale] — 10-point, ordinal scale specifying infant's overall health 5 minutes after birth from 1 (needs immediate medical help) to 10 (in optimal health).
  Units on a Scale | 7 [0 to 9] | 6 [0 to 9] | 6 [0 to 9]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Unfavorable Outcome, Defined as Severe Retinopathy of Prematurity (ROP) or Death Prior to Reaching Acute/Final ROP Status
Description: Death is defined as from any cause before Acute/Final ROP status is determined. ROP was identified by routine ophthalmologic examinations beginning at the latter of 31 weeks PMA or 4-6 weeks chronologic age. The favorable ROP endpoint requires that no ROP, or only mild ROP has occurred in both eyes and the eyes have matured beyond the risk of developing Type 1 ROP (severity meeting criteria for surgical intervention). The unfavorable ROP endpoint requires that one or both eyes reach Type 1 ROP. When ROP did not resolve by the time of discharge, participants were followed as outpatients until reaching an ROP endpoint, up to 55 weeks PMA. Since incomplete follow up is more likely among participants with mild or no ROP than for those with aggressive ROP, an independent adjudication process assigned an ROP endpoint of 'most likely never had Type 1 ROP', or 'most likely developed Type 1 ROP' based on clinical and ROP data review to reduce possible missing data bias.
Time Frame: by 55 weeks PMA
Population: The analysis was performed on an intention to treat basis, including adjudicated ROP endpoints. Individuals for whom adjudicated ROP endpoints could not be obtained were treated as missing completely at random, and excluded from the primary analyses (4 Inositol and 1 Placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Myo-Inositol 5% Injection | 5% Glucose(Dextrose)
Number analyzed (Participants) | 313 | 320
Participants | 91 | 66
Statistical Analysis 1: Comparison: 5% Glucose(Dextrose); The null hypothesis is there is no treatment effect on the development of severe ROP and mortality; Test type: Superiority; p = 0.0095, Robust Poisson — A-priori threshold for statistical significance at 0.05 was specified; Model adjusted for strata defined by center and gestational age; Risk Ratio (RR) = 1.41, 95% CI 2-sided [1.08 to 1.83] — In the risk ratio, the numerator represents the Inositol arm and the denominator represents the placebo arm. (RR>1 implies that the risk of mortality and/or severe ROP is greater in the Inositol group compared to the Placebo group)

2. Secondary Outcome: Number of Participants With Bronchopulmonary Dysplasia (BPD)
Description: BPD is defined as supplemental oxygen required to maintain an oxygenation saturation of >90% at 36 weeks postmenstrual age (PMA) (NICHD physiologic definition).
Time Frame: 36 weeks PMA
Population: The analysis was performed on an intention to treat basis. Individuals for whom BPD outcome could not be obtained were treated as missing completely at random, and excluded from the analyses (45 Inositol and 33 Placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Myo-Inositol 5% Injection | 5% Glucose(Dextrose)
Number analyzed (Participants) | 272 | 288
Participants | 159 | 165
Statistical Analysis 1: Comparison: 5% Glucose(Dextrose); The null hypothesis is there is no treatment effect on the incidence of BPD; Test type: Superiority; p = 0.6599, Robust Poisson regression — A-priori threshold for statistical significance at 0.05 was specified; Model adjusted for strata defined by center and gestational age; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.91 to 1.16] — In the risk ratio, the numerator represents the Inositol arm and the denominator represents the placebo arm. (RR>1 implies that the risk of BPD is greater in the Inositol group compared to the Placebo group)

3. Secondary Outcome: Number of Participants With Bronchopulmonary Dysplasia (BPD) or Death From BPD
Description: BPD is defined as supplemental oxygen required to maintain an oxygenation saturation of >90% at 36 weeks PMA (NICHD physiologic definition). Death from BPD prior to 37 weeks postmenstrual age (PMA) is defined when the cause of death is certified by the Center PI as BPD being the primary cause, or a significant co-contributing cause of death.
Time Frame: prior to 37 weeks PMA
Population: The analysis was performed on an intention to treat basis. Individuals who died prior to 37 weeks PMA for whom the cause(s) of death are unknown or individuals for whom BPD outcome could not be obtained were treated as missing completely at random, and excluded from the analyses (1 Inositol and 5 Placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Myo-Inositol 5% Injection | 5% Glucose(Dextrose)
Number analyzed (Participants) | 316 | 316
Participants | 203 | 195
Statistical Analysis 1: Comparison: 5% Glucose(Dextrose); The null hypothesis is there is no treatment effect on the incidence of BPD or on mortality due to BDP; Test type: Superiority; p = 0.3883, Robust Poisson regression — A-priori threshold for statistical significance at 0.05 was specified; Model adjusted for strata defined by center and gestational age; Risk Ratio (RR) = 1.05, 95% CI 2-sided [0.94 to 1.17]

4. Secondary Outcome: Number of Participants With All Cause Death Before Retinopathy of Prematurity (ROP) Endpoint
Description: Defined as death from any cause following randomization through primary study follow-up (up to 55 weeks postmenstrual age (PMA))
Time Frame: by 55 weeks PMA age
Population: The analysis was performed on an intention to treat basis.
Measure: Count of Participants; unit: Participants
Arm/Group | Myo-Inositol 5% Injection | 5% Glucose(Dextrose)
Number analyzed (Participants) | 317 | 321
Participants | 50 | 33
Statistical Analysis 1: Comparison: 5% Glucose(Dextrose); The null hypothesis is there is no treatment effect on survival to ROP endpoint; Test type: Superiority; p = 0.0306, Robust Poisson regression — A-priori threshold for statistical significance at 0.05 was specified; Model adjusted for strata defined by center and gestational age; Risk Ratio (RR) = 1.53, 95% CI 2-sided [1.03 to 2.25] — In the risk ratio, the numerator represents the Inositol arm and the denominator represents the placebo arm. (RR>1 implies that the risk of mortality prior to ROP endpoint is greater in the Inositol group compared to the Placebo group)

5. Secondary Outcome: Number of Participants With Any Retinopathy of Prematurity (ROP)
Description: ROP was identified by routine ophthalmologic examinations beginning at the latter of 31 weeks PMA or 4-6 weeks chronologic age. Any ROP is defined as ROP of any severity that is observed on at least 2 independent examinations in either eye through the time that Acute/Final ROP status is reached (up to 55 weeks postmenstrual age (PMA)).
Time Frame: by 55 weeks PMA
Population: The analysis was performed on an intention to treat basis. Individuals for whom ROP status could not be defined were treated as missing completely at random, and excluded from the analyses (50 Inositol and 35 Placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Myo-Inositol 5% Injection | 5% Glucose(Dextrose)
Number analyzed (Participants) | 267 | 286
Participants | 171 | 183
Statistical Analysis 1: Comparison: 5% Glucose(Dextrose); The null hypothesis is there is no treatment effect on the incidence of ROP; Test type: Superiority; p = 0.7464, Robust Poisson regression — A-priori threshold for statistical significance at 0.05 was specified; Model adjusted for strata defined by center and gestational age; Risk Ratio (RR) = 1.02, 95% CI 2-sided [0.91 to 1.14]

6. Secondary Outcome: Number of Participants With Type 2 or More Severe Retinopathy of Prematurity (ROP)
Description: Defined as one or both eyes reaching Type 2 ROP (ETROP 2003) or the more severe Type 1 ROP (as defined previously) through the time that Acute/Final ROP status is reached (up to 55 weeks postmenstrual age (PMA)). Type 2 ROP is defined as (ETROP 2003): Stage 3 ROP without Plus Disease (i.e. Zone II) or Stage 1 or 2 ROP without Plus Disease (i.e. Zone I).
Time Frame: by 55 weeks PMA
Population: The analysis was performed on an intention to treat basis. Individuals for whom ROP status and/or type could not be defined were treated as missing completely at random, and excluded from the analyses (54 Inositol and 36 Placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Myo-Inositol 5% Injection | 5% Glucose(Dextrose)
Number analyzed (Participants) | 263 | 285
Participants | 125 | 142
Statistical Analysis 1: Comparison: 5% Glucose(Dextrose); The null hypothesis is there is no treatment effect on the incidence of Type 2 ROP or more severe ROP; Test type: Superiority; p = 0.7598, Robust Poisson regression — A-priori threshold for statistical significance at 0.05 was specified; Model adjusted for strata defined by center and gestational age; Risk Ratio (RR) = 0.98, 95% CI 2-sided [0.83 to 1.14] — In the risk ratio, the numerator represents the Inositol arm and the denominator represents the placebo arm. (RR>1 implies that the risk of Type 2 ROP or more severe ROP is greater in the Inositol group compared to the Placebo group)

7. Secondary Outcome: Number of Participants With Severe Intraventricular Hemorrhage (IVH)
Description: Severe IVH is defined as IVH Grades 3 or 4 on either side of the brain. The evaluation for IVH occurs early (within 28 days from birth) via a cranial sonogram and is classified as described by Papile.
Time Frame: by 28 days PMA
Population: The analysis was performed on an intention to treat basis. Individuals for whom severe IVH status could not be defined were treated as missing completely at random, and excluded from the analyses (6 Inositol and 4 Placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Myo-Inositol 5% Injection | 5% Glucose(Dextrose)
Number analyzed (Participants) | 311 | 317
Participants | 51 | 50
Statistical Analysis 1: Comparison: 5% Glucose(Dextrose); The null hypothesis is there is no treatment effect on the incidence severe IVH; Test type: Superiority; p = 0.8133, Robust Poisson regression — A-priori threshold for statistical significance at 0.05 was specified; Model adjusted for strata defined by center and gestational age; Risk Ratio (RR) = 1.04, 95% CI 2-sided [0.74 to 1.48] — In the risk ratio, the numerator represents the Inositol arm and the denominator represents the placebo arm. (RR>1 implies that the risk of severe IVH is greater in the Inositol group compared to the Placebo group)

8. Other Pre Specified Outcome: The Occurrence of Adverse Events and Serious Adverse Events
Time Frame: 7 days post study drug discontinuation
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Necrotizing Enterocolitis (NEC)
Description: Stage II or worse, whether treated (medically or surgically) and if the infant survived (modified Bell's classification [Walsh 1986]).
Time Frame: NRN infant status, i.e., the first occurring of: discharge home, death, transfer, or 120 days following birth
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Isolated Gastrointestinal Perforation
Description: judged not to be due to NEC
Time Frame: NRN infant status, i.e., the first occurring of: discharge home, death, transfer, or 120 days following birth
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Late Onset Sepsis
Description: culture positive septicemia/bacteremia (≥72 hours of age) treated with antibiotics for ≥ 5 days or died before treatment was completed.
Time Frame: NRN infant status, i.e., the first occurring of: discharge home, death, transfer, or 120 days following birth
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Patent Ductus Arteriosus (PDA)
Description: Occurrence of clinically significant patent ductus arteriosus (PDA), and if received intervention with prostaglandin inhibitors, and/or surgery.
Time Frame: NRN infant status, i.e., the first occurring of: discharge home, death, transfer, or 120 days following birth
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Seizures
Description: Seizures treated with an anticonvulsant for >72 hours
Time Frame: NRN infant status, i.e., the first occurring of: discharge home, death, transfer, or 120 days following birth
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Total Days on Parenteral Nutrition
Description: Total days on parenteral nutrition (including amino acids and/or lipids)
Time Frame: NRN infant status i.e., the first occurring of: discharge home, death, transfer, or 120 days following birth
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Days on Oxygen, Days on Ventilator
Time Frame: NRN infant status i.e., the first occurring of: discharge home, death, transfer, or 120 days following birth
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Hearing Loss
Description: Hearing loss as defined as never passing a hearing screening in one or both ears
Time Frame: NRN infant status i.e., the first occurring of: discharge home, death, transfer, or 120 days following birth
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Neurodevelopment
Description: Neurodevelopment at 22-26 months corrected age (i.e., 22-26 months past due date) using the Bayley Scales of Infant Development III.
Time Frame: 22-26 months corrected age
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Vision Loss
Description: Vision loss as diagnosed by an ophthalmologist as legally blind, and subdivided into "ophthalmic origin", or "not ophthalmic origin" (i.e., cortical blindness is non-ophthalmic in origin and indicates that there is no retinal detachment or other abnormal fundus or ocular finding, except optic atrophy. Such cases will be considered central [neurologic] in origin.)
Time Frame: 22-26 Months Corrected Age
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Hearing Loss
Description: Hearing loss requiring that hearing aids be prescribed.
Time Frame: 22-26 Months Corrected Age
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Cerebral Palsy
Description: Cerebral palsy by severity category (absent/mild/moderate/severe).
Time Frame: 22-26 Months Corrected Age
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Overall Health Status
Description: Overall health status per recall from the parent/guardian (including survival, re-hospitalizations, surgeries, ongoing medications, and chronic illnesses).
Time Frame: 22-26 Months Corrected Age
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events will be recorded from treatment initiation until 7 days after the last dose of study drug, up to the earliest of 34 weeks post-menstrual age (PMA), 10 weeks chronologic age (CA), or discharge.
Description: The at-risk population for all-cause mortality is the intent-to-treat (ITT) population which consists of all randomized participants (317 Inositol 321 Placebo). The at-risk population for serious adverse events and/or other (not including serious) adverse events is the safety-population which consists of all individuals who started treatment (313 Inositol 319 Placebo).
Arm/Group | Myo-Inositol 5% Injection | 5% Glucose(Dextrose)
All-Cause Mortality (participants affected / at risk) | 50/317 | 33/321
Serious Adverse Events (participants affected / at risk) | 113/313 | 105/319
Other Adverse Events (participants affected / at risk) | 291/313 | 298/319
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Myo-Inositol 5% Injection (N=313) | 5% Glucose(Dextrose) (N=319)
PULMONARY AIR LEAK (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 9 (10)
PULMONARY HEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 16 (17)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
RESPIRATORY DETERIORATION (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 11 (11)
CHOLESTASIS (Gastrointestinal disorders) | 9 (9) | 3 (3)
DELAYED GASTRIC EMPTYING (Gastrointestinal disorders) | 1 (1) | 1 (1)
ELEVATED LIVER ENZYMES (Gastrointestinal disorders) | 3 (3) | 0 (0)
EMESIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
NEC (Gastrointestinal disorders) | 19 (20) | 14 (16)
SPONTANEOUS INTESTINAL PERFORATION, WITHOUT NEC (Gastrointestinal disorders) | 15 (17) | 20 (24)
SUPERFICIAL INFECTION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SYSTEMIC INFECTION (Infections and infestations) | 50 (55) | 34 (39)
IVH (Nervous system disorders) | 31 (33) | 30 (32)
SEIZURES (Nervous system disorders) | 1 (1) | 3 (3)
BRADYCARDIA (Cardiac disorders) | 0 (0) | 2 (2)
CONGESTIVE HEART FAILURE (Cardiac disorders) | 0 (0) | 1 (1)
HYPERTENSION (Cardiac disorders) | 0 (0) | 2 (2)
PDA (Cardiac disorders) | 8 (8) | 13 (13)
POOR PERFUSION OR HYPOTENSION (Cardiac disorders) | 23 (24) | 14 (16)
ANEMIA (Blood and lymphatic system disorders) | 14 (15) | 10 (11)
HYPERBILIRUBINEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 5 (5)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 9 (9) | 9 (9)
THROMBOCYTOSIS (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
DIURESIS (Renal and urinary disorders) | 1 (1) | 0 (0)
ELEVATED CREATININE (Renal and urinary disorders) | 3 (3) | 0 (0)
HYPERKALEMIA (Renal and urinary disorders) | 4 (4) | 4 (4)
HEMATURIA (Renal and urinary disorders) | 1 (1) | 1 (1)
OLIGURIA (Renal and urinary disorders) | 11 (13) | 7 (8)
PROTEINURIA (Renal and urinary disorders) | 1 (1) | 0 (0)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 6 (6) | 5 (6)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
SKIN BREAKDOWN (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
HYPOXIC RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
CARDIOPULMONARY ARREST (Cardiac disorders) | 1 (1) | 0 (0)
SKIN CELLULITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PULMONARY VALVE STENOSIS (Cardiac disorders) | 1 (1) | 0 (0)
ADRENAL INSUFFICENCY (Endocrine disorders) | 1 (1) | 1 (1)
COAGULOPATHY (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
ESPHOGEAL PERFORATION (Gastrointestinal disorders) | 3 (3) | 1 (1)
ILEUS (Gastrointestinal disorders) | 1 (1) | 1 (1)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
HEPATIC FAILURE (Hepatobiliary disorders) | 0 (0) | 2 (2)
ACIDOSIS (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPONATREMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
HYPERNATREMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 4 (4) | 2 (2)
COMPARTMENT SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MECONIUM PLUG SYNDROME (Gastrointestinal disorders) | 1 (1) | 0 (0)
THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Myo-Inositol 5% Injection (N=313) | 5% Glucose(Dextrose) (N=319)
ANEMIA (Blood and lymphatic system disorders) | 185 (336) | 202 (379)
HYPERBILIRUBINEMIA (Blood and lymphatic system disorders) | 67 (69) | 56 (63)
NEUTROPENIA (Blood and lymphatic system disorders) | 30 (31) | 30 (36)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 31 (40) | 26 (37)
THROMBOCYTOSIS (Blood and lymphatic system disorders) | 95 (108) | 96 (119)
DIURESIS (Renal and urinary disorders) | 36 (83) | 44 (77)
ELEVATED CREATININE (Renal and urinary disorders) | 17 (26) | 16 (24)
HYPERKALEMIA (Renal and urinary disorders) | 45 (54) | 49 (58)
GLUCOSUIRA (Renal and urinary disorders) | 7 (7) | 2 (3)
HEMATURIA (Renal and urinary disorders) | 14 (16) | 14 (17)
OLIGURIA (Renal and urinary disorders) | 46 (79) | 46 (68)
PROTEINURIA (Renal and urinary disorders) | 14 (17) | 9 (14)
PULMONARY AIR LEAK (Respiratory, thoracic and mediastinal disorders) | 23 (25) | 25 (28)
PULMONARY HEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (8)
RESPIRATORY DETERIORATION (Respiratory, thoracic and mediastinal disorders) | 114 (172) | 120 (171)
CONGESTIVE HEART FAILURE (Cardiac disorders) | 20 (20) | 19 (22)
HYPERTENSION (Cardiac disorders) | 23 (32) | 23 (36)
PDA (Cardiac disorders) | 88 (89) | 87 (87)
POOR PERFUSION OR HYPOTENSION (Cardiac disorders) | 36 (45) | 30 (40)
TACHYCARDIA (Cardiac disorders) | 11 (14) | 9 (16)
CHOLEOSTASIS (Gastrointestinal disorders) | 36 (36) | 26 (26)
DELAYED GASTRIC EMPTYING (Gastrointestinal disorders) | 52 (76) | 46 (95)
DIARRHEA (Gastrointestinal disorders) | 4 (4) | 2 (2)
ELEVATED LIVER ENZYMERS (Gastrointestinal disorders) | 18 (20) | 16 (17)
EMESIS (Gastrointestinal disorders) | 2 (2) | 4 (4)
NEC (Gastrointestinal disorders) | 16 (16) | 14 (14)
SPONTANEOUS INTESTINAL PERFORATION WITHOUT NEC (Gastrointestinal disorders) | 2 (2) | 2 (2)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 78 (97) | 67 (88)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 7 (10) | 10 (10)
LOCAL INFECTION (Infections and infestations) | 10 (10) | 8 (9)
SUPERFICIAL INFECTION (Infections and infestations) | 10 (11) | 18 (18)
SYSTEMIC INFECTION (Infections and infestations) | 76 (98) | 84 (102)
ABNORMAL MOVEMENTS (Nervous system disorders) | 0 (0) | 1 (1)
IVH (Nervous system disorders) | 36 (36) | 33 (33)
SEIZURES (Nervous system disorders) | 8 (8) | 5 (5)
STATE OF ALERTNESS (Nervous system disorders) | 3 (5) | 3 (3)
RASH (Skin and subcutaneous tissue disorders) | 4 (5) | 5 (5)
SKIN BREAKDOWN (Skin and subcutaneous tissue disorders) | 7 (7) | 4 (4)
HYPOTHERMIA (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
OTHER (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Other (not including serious) adverse events under blood and lymphatic system disorders includes frank blood drainage from Penrose drain.
OTHER (Cardiac disorders) | 0 (0) | 2 (2) — Other (not including serious) adverse events under cardiac disorders include atrial vegetation/thrombus, femoral continuous loop complication (under perfusion right leg and great toe)
RENAL DYSFUNCTION (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 1 (1)
BILATERAL HYDRONEPHROSIS (Renal and urinary disorders) | 0 (0) | 1 (1)
CHRONIC LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (7)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
ABDOMINAL DISTENTION (Gastrointestinal disorders) | 0 | 1 (1)
BLOODY STOOL (Gastrointestinal disorders) | 1 (1) | 1 (1)
BOWEL DYSFUNCTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
ESOPHOGEAL PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
FEEDING INTOLERANCE (Gastrointestinal disorders) | 2 (3) | 2 (2)
GASTRITIS (Gastrointestinal disorders) | 1 (1) | 1 (1)
GASTROINTESTINAL FISTULA (Gastrointestinal disorders) | 0 (0) | 2 (2)
ILEUS (Gastrointestinal disorders) | 0 (0) | 1 (1)
STRICTURES REQUIRING SURGERY (Gastrointestinal disorders) | 1 (1) | 0 (0)
ACIDOSIS (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERTHYROIDISM (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOTHYROIDISM (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
ELEVATED 17-OH PROGESTERONE (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
RICKETS (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
HYPONATREMIA (Metabolism and nutrition disorders) | 7 (7) | 5 (5)
HYPERNATREMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERTRIGLYCERIDEMIA (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
IV INFILTRATE (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 0 (0) | 4 (4)
INTRACRANIAL HEMORRHAGE (Nervous system disorders) | 0 (0) | 1 (1)
OSTEOPENIA (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (6)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ATOPIC DERMATITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SOFT TISSUE NECROSIS (UPPER LIMB) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
THROMBOSIS (Vascular disorders) | 2 (2) | 0 (0)
GRANULATION TISSUE PROLAPSE (PENROSE DRAIN SITE) (Gastrointestinal disorders) | 1 (1) | 0 (0)
NASAL SEPTIC BREAKDOWN (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to a manufacturing issue, enrollment and treatment were temporarily suspended pending review of primary outcome data for the enrolled infants. The statistically significant increase in mortality resulted in early study termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators must adhere to the Neonatal Research Network Publication policies.